CLINICAL TRIAL: NCT06324682
Title: Evaluation of conTempoRary Cardiac Stimulation in Clinical practicE: lEft, BivEntriculAr, Right, and conDuction System Pacing
Brief Title: ConTempoRary Cardiac Stimulation in Clinical practicE: lEft, BivEntriculAr, Right, and conDuction System Pacing
Acronym: TREEBEARD
Status: Recruiting | Type: Observational
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Matteo Bertini, Professor, University Hospital of Ferrara
Other Study IDs: 825/2022/Oss/AOUFe
Record Dates: First submitted 2024-01-31; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Arrhythmias, Cardiac; Atrioventricular Block; Reduced Systolic Function; Atrial Fibrillation; Bradyarrhythmia; Ventricular Tachycardia; Ventricular Dysfunction; Ventricular Fibrillation; Ventricular Arrythmia; Atrioventricular Nodal Disease; Atrioventricular Conduction Defects; Atrioventricular Block Complete; Atrioventricular Block Incomplete; Atrioventricular Junctional Rhythm; Bundle-Branch Block; Left Bundle-Branch Block; Heart Failure, Systolic; Block;Atrioventricular; Block; Arrhythmic; Block; Mobitz; Block, Heart; Block, Fascicular; Block Branch Bundle Left; Heart Failure，Congestive; Heart Arrhythmia
Keywords: Pace maker (PM); Implantable cardioverter defibrillator (ICD); Atrioventricular Block; Bradyarrhythmia; Ventricular Dysfunction; Cardiac Resynchronization therapy; Conduction System Pacing; His Pacing; Left bundle branch area pacing (LBBAP); CRT; CSP; Primary prevention; Secondary prevention; Atrioventricular Block Complete; Heart failure; Ventricular Arrythmia; Ventricular Fibrillation; Ventricular Tachycardia
MeSH Terms: conditions — Arrhythmias, Cardiac; Atrioventricular Block; Atrial Fibrillation; Bradycardia; Tachycardia, Ventricular; Ventricular Dysfunction; Ventricular Fibrillation; Bundle-Branch Block; Heart Failure, Systolic; Bites and Stings; Heart Block; Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Conventional right ventricular (RV) pacing: The device (pace maker or implantable cardiac defibrillator) is implanted in the subcutaneous subclavian area (right or left) and it is connected to transvenous lead/leads (active or passive) implanted in the right cardiac chambers (atrium and ventricle or ventricle only), which detect intrinsic electrical activity and stimulate when needed. The ventricle pacing might be obtained with an apical or septal stimulation.
  Vascular access might be from the cephalic, axillary or subclavian veins. Once positioned, lead's pacing threshold, sensing and impedance are measured. If the investigators find good and stable electrical parameters, the catheter(s) is(are) fixed and left in place.
  Interventions: Device: Cardiac pacing - Conventional RV pacing
- Conduction System Pacing: The approach for the insertion of the device and of the transvenous leads is similar to the previous ones.
  The ventricle activation might be obtained with the his bundle stimulation or with the left bundle branch area pacing downstream of the conduction block. Vascular access might be from the cephalic, axillary or subclavian veins.
  Both selective and non-selective stimulation of the His bundle and the stimulation of the left bundle branch and left septum are considered successful. In both cases, attempts are made to locate the atrio-ventricular junction by fluoroscopic methods or with three-dimensional electroanatomical mapping system. The Hisian potential is sought and the catheter is positioned. In the LBBAP the investigators place the lead 1.5 cm below the His region and, with the pacemaking method, the investigators identify an area that electrocardiographically shows a W signal in V1 lead with D2 more positive than D3 - after checking the electrical parameters.
  Interventions: Device: Cardiac pacing - Conduction System Pacing
- Cardiac resynchronization therapy (CRT) either -pacing (CRTP) or -defibrillation (CRTD): The approach for the insertion of the device and of the transvenous leads is similar to the previous ones.
  The right ventricle pacing (with a pacing lead or a defibrillation coil) might be obtained with an apical or septal stimulation, while the left ventricular pacing is achieved by placing a catheter (active or passive) in the posterolateral area through a venous branch of the coronary sinus.
  Cardiac resynchronisation therapy (CRT) delivers biventricular or left ventricular only pacing.
  Vascular access might be from the cephalic, axillary or subclavian veins. Once positioned, lead's pacing threshold, sensing and impedance are measured. If the investigators find good and stable electrical parameters, the catheter(s) is(are) fixed and left in place - paying attention to the phrenic nerve capture threshold.
  Interventions: Device: Cardiac pacing - Cardiac resynchronization therapy (pacing - CRTP - or defibrillation - CRTD)
- Epicardial pacing: The device is usually placed in the subcutaneous abdominal area and the lead(s) is(are) secured in the epicardial surface. It is often used in congenital heart defects or post-cardiac surgery scenarios.
  Surgeons may access the epicardium during open-heart surgery or with minimally invasive techniques.
  Interventions: Device: Cardiac pacing - Epicardial pacing
- Leadless pacing: The leadless device is placed via a percutaneous approach through a large-calibre (femoral) vein inside the right ventricle. It is suitable for patients needing a single chamber pacing such as patients with permanent atrial fibrillation with slow ventricular response, in some cases of paroxysmal atrioventricular block, or patients with a history of CIED infections.
  The only one currently available has a cardiac muscle fixation system consisting of 4 self-expanding barbs.
  Once positioned, pacing threshold, sensing and impedance are measured. If the investigators find good and stable electrical parameters, the catheter is left in place.
  Interventions: Device: Cardiac pacing - Leadless pacing

INTERVENTIONS:
Device: Cardiac pacing - Conventional RV pacing — Implantation of devices for cardiac pacing/defibrillation
  Other Names: Cardiac defibrillation - Conventional RV pacing
  Groups: Conventional right ventricular (RV) pacing
Device: Cardiac pacing - Conduction System Pacing — Implantation of devices for cardiac pacing/defibrillation
  Other Names: Cardiac defibrillation - Conduction System Pacing
  Groups: Conduction System Pacing
Device: Cardiac pacing - Cardiac resynchronization therapy (pacing - CRTP - or defibrillation - CRTD) — Implantation of devices for cardiac pacing/defibrillation
  Other Names: Cardiac defibrillation - Cardiac resynchronization therapy (pacing - CRTP - or defibrillation - CRTD)
  Groups: Cardiac resynchronization therapy (CRT) either -pacing (CRTP) or -defibrillation (CRTD)
Device: Cardiac pacing - Epicardial pacing — Implantation of devices for cardiac pacing/defibrillation
  Other Names: Cardiac defibrillation - Epicardial pacing
  Groups: Epicardial pacing
Device: Cardiac pacing - Leadless pacing — Implantation of devices for cardiac pacing/defibrillation
  Other Names: Cardiac defibrillation - Leadless pacing
  Groups: Leadless pacing

SUMMARY:
The goal of this observational study is to evaluate the clinical characteristics of patients undergoing permanent cardiac pacing and to compare procedural efficacy and safety of different implantation approaches in the clinical practice of the participating centres. The contribution of non-fluoroscopic anatomical and electrophysiological reconstruction systems to device implantation procedures will also be evaluated.

Participants [patients over 18 years old with an indication to receive a definitive pacemaker/intracardiac defibrillator implant] will receive a permanent cardiac pacing implant as requested according to European Society of Cardiology (ESC) guidelines; the investigators will evaluate procedural efficacy and safety of different implantation approaches.

DETAILED DESCRIPTION:
Cardiac pacing with implantable electronic cardiac devices and transvenous leads has been introduced since 1960 and is considered a safe, effective and low-risk therapy. The most common indications for permanent cardiac pacing are sinus node dysfunction and atrioventricular blocks. In Europe, pacemaker implants exceed 1000 per million inhabitants. The aim of this therapy is not only to improve patients survival but also their quality of life, which is an essential aspect in assessing patients clinical status and prognosis.

Nowadays, five types of cardiac pacing are recognised in clinical practice:

* Endocardial right chambers pacing: the device is implanted in the subcutaneous subclavian area and it is connected to transvenous leads implanted in the right cardiac chambers, which detect intrinsic electrical activity and stimulate when needed;
* Epicardial pacing: this procedure is often performed in conjunction with cardiac surgery;
* Cardiac resynchronisation therapy (CRT): it delivers biventricular or left ventricular pacing in order to correct interventricular electromechanical dyssynchrony and to improve cardiac output;
* Conduction system pacing: it stimulates the His bundle or the left bundle branch area downstream of the conduction block, in order to restore a physiological electromechanical activation.
* Leadless pacing: via a percutaneous approach through a large-calibre vein, leadless device is placed inside the right ventricle.

These pacing modalities have different possibilities to restore a normal cardiac electromechanical activation, resulting in different degrees of mechanical efficiency in terms of systolic output and diastolic pressures, with consequent effects on improvement/onset of heart failure and cardiopulmonary performance of our patients.

Right ventricular pacing induces a dyssynchronous cardiac activation pattern that can lead to left systolic dysfunction and a consequent increased risk of death related to the development of heart failure.

These observations led to the study of alternative cardiac pacing modalities since the 1990s, in order to improve the clinical outcome of patients with symptomatic bradyarrhythmias. The study of pathological ventricular activation due to left bundle-branch block represents the pathophysiological premise of cardiac resynchronisation in patients with systolic dysfunctional heart failure, and constitutes the developmental model for physiological pacing.

CRT improves mortality and quality of life in patients with heart failure and reduced left ventricular ejection fraction. Typically left ventricular pacing is achieved by placing a catheter in the posterolateral area through a venous branch of the coronary sinus. Unfortunately, despite several years of experience in this field, clinical non-response to this therapy is observed in between 20% and 40% of patients, mostly due to the inability to reach the appropriate pacing site because of anatomical difficulties/absence of veins in the target area.

Recently, conduction system pacing (CSP) has rapidly emerged as an alternative pacing modality to both right ventricular pacing (RVP) and CRT, in order to achieve a more physiological pacing. His bundle pacing (HBP) is considered the physiological pacing "par excellence", but the results in literature show rather frequent technical difficulties due to high pacing thresholds, inadequate ventricular signal amplitude for the detection of intrinsic cardiac activity, low success rate and risk of progression of conduction system pathology in patients with infranodal conduction defects.

Left bundle area pacing has more recently emerged as a viable alternative to achieve physiological pacing with haemodynamic parameters similar to those of HBP, but with lower and stable pacing thresholds, ventricular signal amplitude adequate for the detection of intrinsic cardiac activity and high success rate.

Several experiences with different pacing systems have been published, mainly single-centre studies with small sample sizes and different definitions of conduction system pacing success.

In non-randomised comparative studies, and thus with methodological limitations, clinical superiority over conventional right ventricular pacing, and a substantial efficacy equivalent to CRT in patients with left bundle-branch block, has been shown, creating the preconditions for widespread use of the CSP.

Considering, therefore, the widespread use of the latter technique and the high rate of implants that can potentially benefit from physiological pacing, evaluating safety, feasibility, timing and benefits becomes more crucial than ever.

Therefore, the goal of this observational study is to evaluate the clinical characteristics of patients undergoing permanent cardiac pacing and to compare procedural efficacy and safety of different implantation approaches in the clinical practice of the participating centres.

The contribution of non-fluoroscopic anatomical and electrophysiological reconstruction systems to device implantation procedures will also be evaluated.

The investigators will collect clinical and procedural data from patients with an indication for permanent cardiac pacing who have consecutively undergone an implantable electronic device implant procedure at the Electrophysiology Laboratories of the participating centres over a period of 120 months from the time of approval with a follow-up of an equal 120 months.

Patients will be classified according to the type of stimulation:

1. Right chambers endocardial pacing;
2. Cardiac resynchronisation therapy;
3. Conduction system pacing:

   1. His bundle pacing
   2. Left bundle branch area pacing. In addition, the efficacy and safety at 30 days, and the efficacy and safety at 6 and 12 months of the various pacing modalities, will be evaluated.

The investigators defined efficacy at 30 days the presence of stable electrical parameters - or, if unstable, not requiring early re-intervention, the absence of cardiovascular hospitalizations and the absence of cardiovascular death.

The investigators defined safety at 30 days the absence of procedural complications, such as haematoma requiring re-intervention or with haemoglobin loss >2gr/dl, pneumothorax, pericardial effusion requiring drainage, lead dislocation, cardiac implantable electronic device (CIED) infection or a re-intervention for any cause.

Equally, the investigators defined efficacy at 6-12 months the presence of stable electrical parameters - or, if unstable, not requiring re-intervention, the absence of cardiovascular hospitalizations, the absence of cardiovascular death, the occurrence of heart failure, the occurrence or worsening of atrial or ventricular tachyarrhythmias.

Therefore, the investigators defined safety at 6-12 months the proper functioning of the device, the absence of infection and the absence of re-intervention for any cause.

ELIGIBILITY:
Inclusion Criteria:

* Indication for cardiac stimulation
* Having performed the implantation of a device for cardiac stimulation

Exclusion Criteria:

* Age < 18 years;
* Pregnancy status;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an indication for permanent cardiac stimulation who have subsequently undergone an implantation procedure for an implantable electronic device at the Electrophysiology Laboratories of participating centers within a period of 120 months from the time of approval, with a corresponding follow-up period of another 120 months.
Sampling Method: Non-Probability Sample
Enrollment: 8400 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2033-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
30 days efficacy | 30 days
  Number of successful implantations, defined as the achievement of the planned pacing modality
Rate of hospitalizations for heart failure at 12 months | 12 months
  The investigators considered the worsening of heart failure requiring hospital management
All cause death at 12 months | 12 months
  The investigators will monitor patient's all causes death

SECONDARY OUTCOMES:
All cause and cardiovascular death at 1, 3, 5, 10 years | 120 months
  The investigators will monitor patient's all causes and cardiovascular death
Onset/worsening of heart failure | 120 months
  The investigators will assess patient's hemodynamic stability over the years, monitoring the onset or the worsening of heart failure
Onset/worsening of atrial tachyarrhythmias | 120 months
  The investigators will monitor patient's rhythm over the years, assessing the onset or the worsening of atrial tachyarrhythmias.
Onset/worsening of ventricular tachyarrhythmias | 120 months
  The investigators will monitor patient's rhythm over the years, assessing the onset or the worsening of ventricular tachyarrhythmias.
Procedural time | implantation procedure
  The investigators will evaluate procedural time of different cardiac pacing modalities
Fluoroscopy time | implantation procedure
  The investigators will evaluate fluoroscopy time of different cardiac pacing modalities
Radiation exposure | implantation procedure
  The investigators will evaluate radiation exposure of different cardiac pacing modalities monitoring the dose area product
Success rate of CRT in heart failure | 120 months
  The investigators consider successful CRT if obtain a left ventricular end-systolic volume reduction >15%
Cardiac perforation rate | 30 days
  The investigators will evaluate how often cardiac perforation occurs in relation to the total number of implants and in the various pacing modalities
Hemothorax rate | 30 days
  The investigators will evaluate how often hemothorax occurs in relation to the total number of implants and in the various pacing modalities
Pneumothorax rate | 30 days
  The investigators will evaluate how often pneumothorax occurs in relation to the total number of implants and in the various pacing modalities
Pocket hematoma rate | 30 days
  The investigators will evaluate how often pocket hematoma occurs in relation to the total number of implants and in the various pacing modalities
Pericardial effusion rate | 30 days
  The investigators will evaluate how often pericardial effusion occurs in relation to the total number of implants and in the various pacing modalities
Lead dislocation rate | 120 months
  The investigators will evaluate how often catheter dislocation occurs in relation to the total number of implants and in the various pacing modalities
Lead fracture rate | 120 months
  The investigators will evaluate how often catheter rupture occurs in relation to the total number of implants and in the various pacing modalities
Cardiac Implantable Electronic Devices infections rate | 120 months
  The investigators will evaluate how often infections occur in relation to the total number of implants and in the various pacing modalities
Reintervention rate | 120 months
  The investigators will evaluate how often reintervention is needed in relation to the total number of implants and in the various pacing modalities

CONTACTS AND LOCATIONS:
Overall Officials: Matteo Bertini, MD, PhD, Principal Investigator — Azienda Ospedaliero Universitaria di Ferrara
Locations (31):
- Italy (31):
  - Azienda Ospedaliero-Universitaria di Ferrara, Ferrara, FE
  - Ospedale San Donato, Arezzo
  - Azienda Ospedaliero-Universitaria S.Orsola-Malpighi Bologna, Bologna
  - spedale Maggiore di Bologna, Bologna
  - Ospedale Bernardino Ramazzini, Carpi
  - Ospedale SS Annunziata, Cento
  - Ospedale Bufalini, Cesena
  - Ospedale San Giuseppe, Empoli
  - Ospedale di Vaio, Fidenza
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Ospedale San Giovanni di Dio, Florence
  - Ospedale Santa Maria Annunziata Bagno a Ripoli, Florence
  - Azienda Ospedaliero-Universitaria "Ospedali Riuniti", Foggia
  - Ospedale Morgagni-Pierantoni, Forlì
  - Ospedale Santa Maria della Misericordia Grosseto, Grosseto
  - Ospedale della Versilia, Lido di Camaiore
  - Ospedali Riuniti di Livorno, Livorno
  - Ospedale San Luca, Lucca
  - Nuovo ospedale Apuano Massa, Massa
  - Azienda Ospedaliero-Universitaria Policlinico di Modena, Modena
  - Ospedale Sant'Agostino Estense Modena Baggiovara, Modena
  - Ospedale Civico, azienda Ospedaliera di Palermo, Palermo
  - Policlinico Paolo Giaccone, Palermo
  - Azienda Ospedaliero-Universitaria Maggiore, Parma
  - Ospedale Guglielmo da Saliceto Piacenza, Piacenza
  - Azienda Ospedaliero-Universitaria pisana Cisanello, Pisa
  - Fondazione Toscana Gabriele Monasterio, Pisa
  - Ospedale Santa Maria delle Croci, Ravenna
  - ASMN Reggio Emilia, Reggio Emilia
  - Ospedale degli Infermi Rimini, Rimini
  - Azienda Ospedaliero-Universitaria Senese, Siena

REFERENCES:
- [Derived] Bertini M, Canovi L, Vitali F, Marcantoni L, Pastore G, Volpicelli M, Munciguerra O, Biffi M, Ziacchi M, Rossi L, Carinci V, Sirugo P, Pastori P, Imberti JF, Pellegrino PL, Guerriero E, Sassone B, Bertagnin E, Coppola G, Malagu M, Balla C, Azzolini G, Zuccari G, Zanon F, Boriani G, Zuin M. Two-year outcomes of left bundle branch area pacing versus traditional right ventricular pacing in middle-aged adults: a registry-based trial. Europace. 2025 Aug 4;27(8):euaf181. doi: 10.1093/europace/euaf181. PMID 40880214
- [Derived] Bertini M, Vitali F, Malagu M, Azzolini G, Clo S, Canovi L, Farina J, Bianchi N, De Raffele M, Bianchi C, De Pietri M, Guidi Colombi G, Micillo M, Melpignano A, Pavasini R, Balla C, Guardigli G, Vijayaraman P, Zuin M. Left Ventricular Mechanical Insights Into Left Bundle Branch Pacing and Left Ventricular Septal Pacing. JACC Clin Electrophysiol. 2025 Aug;11(8):1852-1861. doi: 10.1016/j.jacep.2025.03.037. Epub 2025 May 28. PMID 40439650